CLINICAL TRIAL: NCT06455280
Title: A 12-Month, Open-Label Study Evaluating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Siplizumab as Induction Therapy in Patients With Autoimmune Liver Diseases Undergoing Liver Transplantation (SET-SAIL)
Brief Title: A Study of SIPLIZUMAB in AILD and LT Patients
Acronym: SET-SAIL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Elizabeth C. Verna (Other)
Collaborators: ITB-Med LLC (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth C. Verna, Frank Cardile Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU7303
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Liver Disease; Liver Transplant Disorder; Autoimmune Hepatitis; Primary Sclerosing Cholangitis; End Stage Liver DIsease; Cirrhosis, Liver
Keywords: Autoimmune Liver Disease; Liver Transplant Disorder; Autoimmune Hepatitis; Primary Sclerosing Cholangitis; End Stage Liver DIsease; Cirrhosis, Liver
MeSH Terms: conditions — Hepatitis, Autoimmune; Cholangitis, Sclerosing; End Stage Liver Disease; Liver Cirrhosis | interventions — siplizumab

STUDY DESIGN:
Intervention Model Description: Open-Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): subjects will receive 0.6 mg/kg/dose intravenously on the day of transplant (Day 0) intraoperatively and on post-transplant Day 4.
  Interventions: Drug: Siplizumab

INTERVENTIONS:
Drug: Siplizumab — Siplizumab is an anti-CD2 monoclonal antibody that has demonstrated a favorable safety profile of siplizumab in over 779 human subjects and has been shown to target memory T cells-a key driver in the immune processes surrounding rejection and autoimmunity post LT in AILD.

SUMMARY:
There is a significant unmet need for safe and effective therapeutic approaches to prevent immune-mediated graft injury and its complications in liver transplant (LT) recipients with autoimmune liver disease (AILD) including autoimmune hepatitis and primary sclerosing cholangitis. Siplizumab is an anti-cluster of differentiation 2 (CD2) monoclonal antibody that has demonstrated a favorable safety profile of siplizumab in over 779 human subjects and has been shown to target memory T cells-a key driver in the immune processes surrounding rejection and autoimmunity post LT in AILD. The purpose of this pilot, open-label phase 1 study is to determine the safety of siplizumab for induction in patients with AILD undergoing LT.

Up to eight (8) subjects will receive siplizumab 0.6 mg/kg/dose on the day of transplant (Day 0) and Day 4 post-transplant, for a total of two doses.

All subjects will be followed in the study for 12 months post-LT.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety of siplizumab when used as induction immunosuppression in patients with primary sclerosing cholangitis (PSC) or autoimmune hepatitis (AIH) undergoing liver transplantation. Induction immunosuppression drugs are very potent anti-rejection drugs that are given immediately after transplantation to prevent rejection. Siplizumab is investigational, meaning it has not yet been approved for market use for this disease condition by the United States Food and Drug Administration (FDA).

Adult patients (18 years of age and older) listed for LT with the specific AILD diagnoses of PSC or AIH

All subjects will receive 0.6 mg/kg/dose intravenously on the day of transplant (Day 0) intraoperatively and on post-transplant Day 4.

Participation in this study will last approximately 15 months (~ 3 months on the LT waitlist, up to 12 months participation post-LT)

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Age ≥ 18 years old
3. Clinical diagnosis of AIH and/or PSC
4. Listed for liver transplantation
5. Epstein-Barr virus (EBV) seropositive within 12 months of screening

Exclusion Criteria:

1. Presence or history of significant liver disease other than AIH or PSC, including viral hepatitis, alcohol-related liver disease and biopsy-proven non-alcoholic steatohepatitis
2. Prior transplant
3. Listed for multiorgan transplant
4. Acute liver failure
5. Known malignancy, including cholangiocarcinoma and hepatocellular carcinoma
6. Other investigational products in the last 30 days or 5 half lives
7. Pregnant/lactating or unwilling to use contraception
8. Leukopenia (WBC less than 2,000/mm3
9. Absolute lymphocyte count < 200/mm3
10. Sero-positive for HIV-1
11. Hepatitis C Virus (HCV) antibody or RNA positive (within 6 months of screening)
12. HBsAg, hepatitis B virus (HBV) DNA or HBcAb positive (within 6 months of screening)
13. Alcohol use exceeding 30g/day for men or 20g/day for women, and/or known phosphatidylethanol (PETH) level >80 in the 3 months prior to LT
14. Untreated latent TB infection as detected by QuantiFERON Gold Plus Interferon Gamma Release Assay (IGRA) (or current standard interferon gamma release assay for TB)
15. Receipt of any live-attenuated vaccine within 2 months of transplant.

ADDITIONAL exclusion criteria to be reviewed at the time of transplant

1. Renal failure with dialysis or with estimated glomerular filtration rate (eGFR) < 30 at the time of LT
2. Model for end-stage liver disease (MELD)-Na score >30
3. Donor features of Donation after Cardiac Death (DCD), HCV Ab or nucleic acid testing (NAT+), HBcAb or HBsAg+, or blood types A, B, and O incompatible organ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Serious infection in the first month post-transplant, | 1 Month post-transplant
  viral, bacterial or fungal infection that leads to readmission, prolonged hospitalization, reoperation, intensive care unit admission, graft loss or death.

SECONDARY OUTCOMES:
Incidence of immune-mediated liver injury | 12 month Post-transplant
  biopsy proven acute rejection (BPAR), or recurrent AILD
Incidence of graft loss or death | 12 month Post-transplant
  Loss of liver allograft or incidence of mortality
Incidence of BPAR | 12 month Post-transplant
  biopsy proven acute rejection within 12 Month post-transplant
Incidence of treated BPAR | 12 month Post-transplant
  biopsy proven acute rejection that requires treatment within 12 Month post-transplant
Incidence of refractory BPAR | 12 month Post-transplant
  biopsy proven acute rejection within 12 Month post-transplant that is not responsive to treatment
Incidence of development of donor specific antibodies (DSA) | 12 month Post-transplant
  Donor specific antibodies within 12 Month Post-transplant
Incidence of recurrent AILD | 12 month Post-transplant
  based upon histology for autoimmune hepatitis [AIH] and histology and/or imaging for primary sclerosing cholangitis [PSC]

OTHER OUTCOMES:
Peak plasma concentration (Cmax) after single dose of siplizumab | 12 hours Post-treatment
  Cmax after single dose
The area under the curve (AUC) from time zero to the last measurable plasma concentration sampling time. | 84 Days Post-transplant
  AUC based on plasma concentrations over 84 days post-treatment
Descriptive summary statistics by dosing level and visit/sampling time point | 12 month Post-transplant
  the frequency of siplizumab concentrations below the lower-limit of quantification (LLOQ)
Summary statistics of pharmacokinetic (PK) of Siplizumab | 12 month Post-transplant
  mean, standard deviation (SD), coefficient of variation (CV), median, minimum and maximum of siplizumab concentrations.
Change in Concentration T-Cells | 12 month Post treatment
  Change in Concentration of T- cells (cells/uL)
Change in Concentration of B- cells | 12 month Post treatment
  Change in Concentration of B- cells (cells/uL)
Change in Concentration of NK- cells | 12 month Post treatment
  Change in Concentration of NK- cells (cells/uL)
CD2 receptor occupancy by dose level and subject | 12 month Post-transplant
  Measurement of CD2 receptor occupancy
Dynamics of T-cell subset recovery in the blood and allograft liver | 12 month Post-transplant
  Measurement of T-cell subset in the blood and allograft liver

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Verna, MD, Principal Investigator — Columbia University Irving Medical Center/ New York Presbyterian Hospital
Locations (1):
- Columbia University Irving Medical Center/NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: kwong, A., et al., OPTN/SRTR 2018 Annual Data Report: Liver. Am J Transplant, 2020. 20 Suppl s1: p. 193- 299. — https://pubmed.ncbi.nlm.nih.gov/31898413/
- See also: Qian, J., et al., Studies on the induction of tolerance to alloantigens. I. The abrogation of potentials for delayed-type-hypersensitivity response to alloantigens by portal venous inoculation with allogeneic cells. J Immunol, 1985. 134(6): p. 3656-61. — https://pubmed.ncbi.nlm.nih.gov/2580893/
- See also: gugenheim, J., et al., Delayed rejection of heart allografts in hypersensitized rats by extracorporeal donorspecific liver hemoperfusion. Transplantation, 1986. 41(3): p. 398-400. — https://pubmed.ncbi.nlm.nih.gov/3513399/